CLINICAL TRIAL: NCT00235014
Title: A Two-Phase Study for Primary and Secondary Prevention of Diabetic Nephropathy by Combined ACE Inhibition and Calcium Channel Blockade (BENEDICT)
Brief Title: A Study for Prevention of Kidney Disease in Diabetic Patients (BENEDICT)
Acronym: BENEDICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Udo Legler, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VeraTran 083
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension; Diabetes
Keywords: hypertension; diabetes; trandolapril; verapamil; albuminuria
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Albuminuria | interventions — trandolapril; Verapamil; sabadilla

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A-1, B-1 (Active Comparator): A-1 pertains to Phase 1; B-1 pertains to Phase 2
  Interventions: Drug: trandolapril
- A-2, B-2 (Active Comparator): A2 pertains to Phase 1; B-2 pertains to Phase 2
  Interventions: Drug: trandolapril/verapamil
- A-3 (Placebo Comparator)
  Interventions: Drug: placebo
- A-4 (Active Comparator)
  Interventions: Drug: verapamil

INTERVENTIONS:
Drug: trandolapril — 2 mg QD
  Other Names: ABT-878; Mavik/Gopten
  Arms: A-1, B-1
Drug: trandolapril/verapamil — 180/2 mg QD
  Other Names: ABT-TARKA; VeraTran; Tarka
  Arms: A-2, B-2
Drug: placebo — 1 tablet QD
  Arms: A-3
Drug: verapamil — SR 240 mg QD
  Other Names: ABT-150
  Arms: A-4

SUMMARY:
The BENEDICT study is conducted to examine the effects of an ACE inhibitor, calcium channel blockade, a combination of these, and placebo, in the prevention of micro- and macro-albuminuria in Type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Hypertension

Exclusion Criteria:

* Albuminuria (Phase A)
* Non-diabetic renal disease
* Subject has a hypersensitivity to ACE inhibitor, CCB

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Actual)
Dates: Start 1997-03; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Phase A: microalbuminuria; Phase B: progression from microalbuminuria to macroalbuminuria. | 3 years

SECONDARY OUTCOMES:
Course of albumin excretion over time, GFR, blood pressure (BP), incidence of major CV events, overall and CV mortality, HbA1c, progression of retinal changes. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott

REFERENCES:
- [Derived] Rurali E, Noris M, Chianca A, Donadelli R, Banterla F, Galbusera M, Gherardi G, Gastoldi S, Parvanova A, Iliev I, Bossi A, Haefliger C, Trevisan R, Remuzzi G, Ruggenenti P; BENEDICT Study Group. ADAMTS13 predicts renal and cardiovascular events in type 2 diabetic patients and response to therapy. Diabetes. 2013 Oct;62(10):3599-609. doi: 10.2337/db13-0530. Epub 2013 Jun 3. PMID 23733198
- [Derived] Ruggenenti P, Porrini EL, Gaspari F, Motterlini N, Cannata A, Carrara F, Cella C, Ferrari S, Stucchi N, Parvanova A, Iliev I, Dodesini AR, Trevisan R, Bossi A, Zaletel J, Remuzzi G; GFR Study Investigators. Glomerular hyperfiltration and renal disease progression in type 2 diabetes. Diabetes Care. 2012 Oct;35(10):2061-8. doi: 10.2337/dc11-2189. Epub 2012 Jul 6. PMID 22773704
- [Derived] Ruggenenti P, Fassi A, Ilieva A, Iliev IP, Chiurchiu C, Rubis N, Gherardi G, Ene-Iordache B, Gaspari F, Perna A, Cravedi P, Bossi A, Trevisan R, Motterlini N, Remuzzi G; BENEDICT-B Study Investigators. Effects of verapamil added-on trandolapril therapy in hypertensive type 2 diabetes patients with microalbuminuria: the BENEDICT-B randomized trial. J Hypertens. 2011 Feb;29(2):207-16. doi: 10.1097/hjh.0b013e32834069bd. PMID 21243736
- [Derived] Ruggenenti P, Iliev I, Costa GM, Parvanova A, Perna A, Giuliano GA, Motterlini N, Ene-Iordache B, Remuzzi G; Bergamo Nephrologic Diabetes Complications Trial Study Group. Preventing left ventricular hypertrophy by ACE inhibition in hypertensive patients with type 2 diabetes: a prespecified analysis of the Bergamo Nephrologic Diabetes Complications Trial (BENEDICT). Diabetes Care. 2008 Aug;31(8):1629-34. doi: 10.2337/dc08-0371. Epub 2008 Apr 28. PMID 18443191